CLINICAL TRIAL: NCT00058331
Title: A Phase III, Randomized Study Of Two Different Dosing Schedules Of Erythropoetin In Anemic Patients With Cancer
Brief Title: Epoetin Alfa in Treating Anemia in Patients With Solid Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCCTG-N02C2; CDR0000288821 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Anemia; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Anemia; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- epoetin alfa - long term dosing (Experimental): Patients receive epoetin alfa (EPO) subcutaneously (SC) once weekly for 3 weeks. Then patients receive EPO SC once weekly for 18 weeks. Quality of life is assessed at randomization at then monthly during study treatment.
  Patients are followed every 6 months for 1 year.
  Interventions: Biological: epoetin alfa
- epoetin alfa - short term dosing (Experimental): Patients receive epoetin alfa (EPO) subcutaneously (SC) once weekly for 3 weeks. Patients receive EPO SC on day 1 of weeks 4, 7, 10, 13, 16, and 19. Quality of life is assessed at randomization at then monthly during study treatment.
  Patients are followed every 6 months for 1 year.
  Interventions: Biological: epoetin alfa

INTERVENTIONS:
Biological: epoetin alfa

SUMMARY:
RATIONALE: Epoetin alfa may stimulate red blood cell production and treat anemia in patients with solid tumors. It is not yet known whether epoetin alfa given once a week is more effective than epoetin alfa given once every 3 weeks in treating anemia.

PURPOSE: Randomized phase III trial to study the effectiveness of epoetin alfa in treating anemia in patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effects of 2 different schedules of epoetin alfa on decreasing transfusion requirements in anemic patients with nonmyeloid cancer.
* Compare the effects of these regimens on increasing hemoglobin levels in these patients.
* Compare the effects of these regimens on overall quality of life (QOL) and anemia-specific components of QOL in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to concurrent chemotherapy or radiotherapy (yes vs no), concurrent platinum-based (cisplatin or carboplatin) chemotherapy (yes vs no), degree of anemia (mild [hemoglobin at least 9.0 g/dL] vs severe [hemoglobin less than 9.0 g/dL]), age (60 and under vs over 60), and type of neoplasm (plasma cell disorder [including multiple myeloma] or lymphoproliferative disorder [including non-Hodgkin's lymphoma and chronic lymphocytic leukemia] vs all other neoplasms).

All patients receive epoetin alfa (EPO) subcutaneously (SC) once weekly for 3 weeks. Patients are then randomized to 1 of 2 treatment arms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a nonmyeloid cancer (excluding nonmelanoma skin cancer)
* Anemia secondary to cancer or cancer treatment*

  * Hemoglobin less than 12 g/dL (males)
  * Hemoglobin less than 11 g/dL (females) NOTE: *Active anticancer therapy is not required for study enrollment
* Anemia must not be secondary to any of the following:

  * B_12, folic acid, or iron deficiency

    * Ferritin must be normal or elevated
  * Gastrointestinal bleeding or hemolysis
  * Primary or chemotherapy-induced myelodysplastic syndromes
* No untreated CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 6 months

Cardiovascular

* No history of uncontrolled cardiac arrhythmias
* No history of deep venous thrombosis within the past year (unless on anticoagulation)
* No uncontrolled hypertension (systolic blood pressure at least 180 mm Hg and diastolic blood pressure at least 100 mm Hg) within the past year (unless on anticoagulation)

Pulmonary

* No history of pulmonary embolism within the past year (unless on anticoagulation)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No known hypersensitivity to epoetin alfa, mammalian cell-derived products, or human albumin
* No new onset of seizures within the past 3 months
* No poorly controlled seizures
* Able and willing to complete quality of life forms
* Alert and mentally competent to give informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 6 months since prior epoetin alfa
* More than 6 months since any prior investigational forms of epoetin alfa (e.g., gene-activated epoetin alfa or novel erythropoiesis-stimulating protein)
* No concurrent peripheral blood stem cell transplantation
* No concurrent bone marrow transplantation

Surgery

* More than 14 days since prior major surgery

Other

* More than 2 weeks since prior red blood cell transfusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2003-06; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Compare the effects of these regimens on increasing hemoglobin levels | Up to 1 year post-treatment

SECONDARY OUTCOMES:
Compare the effects of these regimens on overall quality of life (QOL) | Up to 1 year post-treatment
Compare the effects of anemia-specific components of QOL | Up to 1 year post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: David P. Steensma, MD, Study Chair — Dana-Farber Cancer Institute
Locations (18):
- United States (18):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Steensma DP, Molina R, Sloan JA, Nikcevich DA, Schaefer PL, Rowland KM Jr, Dentchev T, Novotny PJ, Tschetter LK, Alberts SR, Hogan TF, Law A, Loprinzi CL. Phase III study of two different dosing schedules of erythropoietin in anemic patients with cancer. J Clin Oncol. 2006 Mar 1;24(7):1079-89. doi: 10.1200/JCO.2005.02.7276. PMID 16505427
- [Result] Steensma DP, Molina R, Sloan JA, et al.: A phase III randomized trial of two different dosing schedules of erythropoietin (EPO) in patients with cancer-associated anemia: North Central Cancer Treatment Group (NCCTG) study N02C2. [Abstract] J Clin Oncol 23 (Suppl 16): A-8031, 736s, 2005.